CLINICAL TRIAL: NCT07316725
Title: the Effect of Virtual Reality Exercise on Selected Electrolytes Levels in Intradialytic Patients
Acronym: VRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, sarah mostafa mohamed, principle investigator : sarah mostafa mohamed, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005982
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Diseases
Keywords: Virtual Reality Exercise; Selected Electrolytes Levels; Intradialytic Patients
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Exergaming; Standard of Care

STUDY DESIGN:
Intervention Model Description: virtual reality and standard care
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Exercise (Experimental): Twenty patients will receive virtual reality exercise during dialysis sessions three times per weeks for 3 months (30 minutes of guided VR exercise).
  Interventions: Other: Virtual Reality Exercise; Other: standard care
- standard care (Active Comparator): Twenty patients will receive standard care during dialysis sessions three times per weeks for 3 months.
  Interventions: Other: standard care

INTERVENTIONS:
Other: Virtual Reality Exercise — the patients will receive 30 minutes virtual reality exercise; (5 minutes warm Up stretching exercise - 20 minutes cycling exercise -5 minutes cool down stretching exercise) plus standard care
  Arms: Virtual Reality Exercise
Other: standard care — the patients will receive standard care in the form of medical care

SUMMARY:
this study will be conducted to investigate the effect of Intra-Dialysis virtual reality exercise on selected electrolytes balance in patients with end stage renal disease.

DETAILED DESCRIPTION:
Chronic Kidney Disease (CKD) is a progressive condition that often leads to end-stage renal disease, requiring dialysis. Patients undergoing hemodialysis frequently experience physical inactivity and electrolyte imbalances, which can adversely affect their health outcomes. Regular physical activity is crucial for maintaining muscle strength and physical function in CKD patients.Electrolytes play vital roles in various physiological functions, including muscle contraction, nerve transmission, and fluid balance. In end stage renal disease patients, imbalances can lead to serious complications, including: hyperkalemia, Hyponatremia, and hypocalcemia.VR has been employed in medicine to assist patients in recovering their motor and cognitive abilities. It has proven effective in enhancing physical functions such as posture, balance, and motor skills. When combined with physical exercise, VR has been shown to improve the functional abilities and quality of life of hemodialysis patients. For those with end stage renal disease patients, who experience discomfort during hemodialysis, VR offers a distraction that can reduce the perception of pain, fatigue, nausea, lightheadedness, and headaches, thereby facilitating smoother exercise continuity and enhancing overall adherence to rehabilitation activities. so this study will be conducted to assess the effect of Intra-Dialysis Virtual Reality Exercise on Selected Electrolytes Balance in Patients with End Stage Renal Disease

ELIGIBILITY:
Inclusion Criteria:

* Patients are diagnosed with end stage renal disease on regular dialysis.
* Their ages will be arranged from 20-40 years old.
* All patients are under medical control.
* Patients on regular dialysis more than 3 months.

Exclusion Criteria:

* Visual impairment.
* Severe cognitive impairment.
* Recent major surgery.
* Patients with sever musculoskeletal problems.
* Severe cardiovascular disease limiting exercise.
* Patients with Hemoglobin drop less than 9 g/dl

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Serum Electrolyte Levels | up to three months
  Measurements the level of sodium, potassium, calcium and phosphorus by venous blood sample. the normal value for Sodium: 135-145 mEq/L
  ,Potassium: 3.5-5.0 mEq/L, Calcium: 8.5-10.2 mg/dL, and Phosphorus: 2.5-4.5 mg/dL

SECONDARY OUTCOMES:
blood pressure | up to three months
  A sphygmomanometer will be used to assess blood pressure with normal range 120/80
oxygen saturation levels | up to three months
  A pulse oximeter will be used to assess oxygen saturation level. 95-100% considered normal for healthy individuals
functional exercise capacity | up to three months
  6-Minute Walk Test will be used to assess functional exercises capacity
exercise intensity | up to three months
  The Rated Perceived Exertion (RPE) Scale will be used to assess exercise intensity. it is a subjective 6-20 scale measuring exercise intensity, where 6 is no effort (rest) and 20 is maximum effort.